CLINICAL TRIAL: NCT06838364
Title: Comparison of the Effectiveness of Ultrasound-guided Techniques and Infrared Illumination, Compared With the Standard Approach to Peripheral Venous Line Placement in People With Difficult Venous Access
Acronym: REUSSIR-VVP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REUSSIR-VVP
Record Dates: First submitted 2025-01-07; First posted 2025-02-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Venous Catheterization
Keywords: ultrasound guided; infrared; A-DIVA scale

STUDY DESIGN:
Intervention Model Description: This is a comparative, prospective, controlled, randomized trial with three parallel arms, conducted at a single center, with a superiority design, in patients with difficult venous access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Landmark technique (Active Comparator): The gold standard technique, with observationnal and palpation
  Interventions: Other: Landmark technique
- Infrared peripheral venous technique (Active Comparator): use an infrared device for venous peripheral visualisation and catheter insertion
  Interventions: Other: Infrared peripheral venous technique
- Ultrasound-guided peripheral venous technique (Active Comparator): Use the Ultrasound-guided technique for venous peripheral visualisation and catheter insertion
  Interventions: Other: Ultrasound-guided peripheral venous technique

INTERVENTIONS:
Other: Infrared peripheral venous technique — use a infrared device for venous peripheral visualisation and catheter insertion
  Other Names: 2
  Arms: Infrared peripheral venous technique
Other: Ultrasound-guided peripheral venous technique — Use the ultrasound-guided technique for venous peripheral visualisation and catheter insertion
  Other Names: 1
  Arms: Ultrasound-guided peripheral venous technique
Other: Landmark technique — the gold standard technique with observationnal and palpation
  Other Names: control
  Arms: Landmark technique

SUMMARY:
Introduction

Peripheral venous catheterization (PVC) is the most common invasive procedure in healthcare worldwide. Improving the success rate of PVC on the first attempt is crucial for patients, as it impacts pain, anxiety, the risk of extravasation, rapid access to care, and the patient-provider relationship. For healthcare providers, a higher success rate enhances self-confidence and autonomy, while institutions benefit from improved reputation and reduced costs.

In the Poitiers hosptial, one in ten catheters is used in imaging services, with CT scan departments accounting for 66.3% of catheter usage due to iodinated contrast injections. Literature suggests two techniques to enhance PVC success: ultrasound-guided and infrared illumination methods. These techniques appear effective primarily for patients with difficult venous access. Additionally, the A-DIVA clinical score has been developed to predict first-attempt success rates. However, no studies in Europe have compared the effectiveness of these two techniques in imaging settings or based on the A-DIVA score. This study aims to identify the most effective technique for PVC in patients with difficult venous access.

Objectives

Compare the proportion of successful PVCs on the first attempt among the classical method (Gold Standard), ultrasound-guided technique, and infrared illumination technique in adult patients with difficult venous access.

Compare the proportion of successful PVCs on the second attempt (if the first attempt fails) among the three techniques.

Compare the total number of attempts required for successful PVC. Evaluate the maximum pain experienced by patients during successful PVC. Assess overall patient satisfaction following successful PVC. Evaluate operator satisfaction with the procedure. Measure the time taken for catheterization from material preparation to successful catheter placement.

Analyze the fallback strategies chosen by operators after a failed attempt (e.g., calling a colleague, continuing with the classical method, using ultrasound guidance, infrared illumination, or abandoning the procedure).

Describe the catheter sizes chosen by operators based on the A-DIVA score and the number of failed attempts.

Methodology

This is a prospective, controlled, randomized, three-arm, single-center, superiority trial involving patients with difficult venous access. Inclusion criteria include:

Patients aged 18 years or older. Patients scheduled for a CT scan requiring PVC. Patients with an A-DIVA score of 2 or higher. Patients capable and willing to comply with study procedures. Patients covered by social security or through a third party. Patients providing written informed consent after receiving clear information about the study.

Exclusion criteria include:

Patients with contraindications for PVC (e.g., presence of an arteriovenous fistula, orthopedic or vascular prosthesis, history of mastectomy, etc.).

Patients with contraindications for iodinated contrast injection as defined by the French Society of Radiology.

Patients already included in the study. Vulnerable populations (e.g., minors, pregnant or breastfeeding women, individuals deprived of liberty).

Intervention Groups

Control: Classical method based on clinical examination (visualization and palpation).

Experimental: Ultrasound-guided method. Experimental: Infrared illumination method. Sample Size and Duration

A total of 249 patients will be enrolled, with 82 patients in each group. The inclusion period will last 12 months, and each participant will be involved for a maximum of 4 hours. The total duration of the clinical investigation will be 1 year and 4 hours.

Outcome Measures

The primary outcome is the proportion of successful PVCs on the first attempt, defined as the administration of 5 ml of NaCl without reported pain or visible edema.

The total number of skin penetrations by the catheter will be recorded. Maximum pain will be assessed using a numerical rating scale (0-10). Patient satisfaction will be measured using a similar numerical scale. Operator satisfaction will also be evaluated on a scale from 0 (very dissatisfied) to 10 (very satisfied).

Time for catheterization will be recorded in minutes, starting from the preparation of the PVC tray until successful catheter placement.

The fallback strategy after a failed attempt will be documented. The size of the catheter chosen for each attempt will be recorded. Statistical Analysis

The primary outcome will be compared among the three groups using ANOVA, followed by pairwise comparisons using Tukey's test if significant differences are found.

Expected Outcomes

Identifying the most effective PVC technique could increase the likelihood of first-attempt success in adults with difficult venous access.

Benefits for Patients

Reduced pain and discomfort from multiple attempts. Decreased risk of infection and extravasation. Maintenance of venous integrity. Sustained trust in the patient-provider relationship.

DETAILED DESCRIPTION:
Peripheral venous catheterization (PVC) is the most common invasive medical procedure performed worldwide. Improving the success rate of PVC on the first attempt is crucial for patients in terms of pain, anxiety, risk of extravasation, rapid access to care, maintenance of the patient-caregiver relationship, and for caregivers in terms of self-confidence and autonomy, and for institutions in terms of image and societal cost.

One in ten catheters used in the Territorial Hospital Group of Vienne is used in imaging services, according to the 2021-2022 estimate. Particularly, the scanner services account for 66.3% of catheters ordered in imaging, in relation to the injection of iodinated contrast agent.

The literature presents two techniques that can improve the success rate of PVC, namely ultrasound-guided and infrared illumination methods. Their use appears to be effective only in patients with difficult venous access.

Furthermore, the prediction of the success rate on the first attempt has been made possible thanks to the A-DIVA clinical score. No study has compared the effectiveness of these two techniques in Europe, in imaging, or based on this clinical score. The objective of the study is to determine the most effective technique for successful PVC in patients with difficult venous access.

Compare the proportion of successful peripheral venous catheterizations on the first attempt between the classical method (Gold Standard), ultrasound-guided technique, and infrared illumination technique in adult patients with difficult venous access.

Catheterization is defined as the successful administration of 5 ml of NaCl without pain expressed by the patient or visible edema (absence of diffusion or hematoma) immediately after the first skin puncture by the catheter.

The primary outcome measure is binary and evaluated on the first attempt.

Compare the proportion of successful peripheral venous catheterizations on the second attempt (if the first attempt fails) between the classical method (Gold Standard), ultrasound-guided technique, and infrared illumination technique in adult patients with difficult venous access.

Compare the total number of attempts Evaluate the maximum pain experienced by the patient when PVC is successful Evaluate the patient's overall satisfaction when PVC is successful Evaluate the operator's overall satisfaction Time required for catheterization from the end of material preparation to successful catheterization.

Analyze the recourse system chosen by the caregiver after a first failure (calling a colleague, continuing with the classical method, ultrasound-guided technique, infrared illumination technique, or abandoning PVC).

Describe the catheter calibers chosen by caregivers based on the A-DIVA score and the number of failed attempts.

The success of catheterization is defined as the absence of pain expressed by the patient, or visible edema downstream of the perfusion site (absence of diffusion or hematoma) after the administration of 5 ml of NaCl, during the second skin puncture by the catheter (1 puncture = 1 attempt).

Total number of skin punctures by a catheter. The maximum pain will be evaluated using a numerical scale from 0 to 10. This scale is sensitive, reproducible, reliable, and widely used in scientific literature. The evaluation will follow the question "On a scale of 0 to 10, with 0 being no pain and 10 being the maximum imaginable pain, how would you rate the maximum pain you experienced during your perfusion?" The patient's satisfaction will be measured using a numerical scale by answering the question "On a scale of 0 to 10, with 0 being very dissatisfied and 10 being completely satisfied, how would you rate your overall satisfaction with your perfusion?" The operator's satisfaction will be evaluated using a numerical scale from 0 (very dissatisfied) to 10 (completely satisfied) by answering the question "Are you satisfied with the placement of this catheter?" The time will be recorded in minutes, starting after the preparation of the PVC tray by the operator. This includes vein location, skin disinfection, tourniquet placement, catheterization, connection to the perfusion line, securing with bandages, and occlusive dressing. If a failure is observed, the timer will not be stopped, and the time will be recorded until vascular access is obtained, including the time required for alternative procedures.

In case of failure, indicate the success or need for recourse for the caregiver. The type of recourse chosen will be recorded: calling a colleague, continuing with the classical method, ultrasound-guided technique, infrared illumination technique, or abandoning PVC.

For each attempt, describe the catheter caliber chosen: 14 Ga (Orange) / 16 Ga (Gray) / 18 Ga (Green) / 20 Ga (Pink) / 22 Ga (Blue) / 24 Ga (Yellow) / 26 Ga (Purple) This is a comparative, prospective, controlled, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Patient with a CT scan appointment and a medical prescription requiring a peripheral venous line.
* Patient with an A-DIVA score greater than or equal to 2.
* Patient able and willing to comply with all study procedures.
* Patient covered by a social security scheme or covered through a third party.
* Patients who have given their free and informed written consent following clear and fair information about the study.

Exclusion Criteria:

* Patient with a contraindication to VVP insertion:
* Arm with arteriovenous fistula
* Limb with an orthopaedic or vascular prosthesis
* Previous mastectomy, axillary lymph node dissection or homolateral radiotherapy of the arm
* Paralysed limb
* Presence of haematomas or puncture site wounds
* Limb with phlebitis or infection
* Patients already included in the study
* Persons benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, pregnant or breast-feeding women, adults under legal protection and patients in emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the success of catheterization | Up to 4 hours
  Absence of pain expressed by the patient, or visible oedema (absence of signs of diffusion or haematoma)

SECONDARY OUTCOMES:
Evaluate the Success of catheterisation | Up to 4 hours
  Absence of pain expressed by the patient, or visible oedema (absence of signs of diffusion or haematoma)
Evaluate the number of attempts | Up to 4 hours
  Compare the total number of attempts
Evaluate the maximum pain felt by the patient when the peripheral venous insertion is successfully inserted. | Up to 4 hours
  A lickert scale from 0 to 10. Lower mean a worst outcome.
Evaluate patient satisfaction | Up to 4 hours
  A lickert scale from 0 to 10. Lower scores mean a worst outcome.
Evaluate overall care giver satisfaction | Up to 4 hours
  A lickert scale from 0 to 10. Lower scores mean a better response.
Evaluate the cathetrization time | Up to 4 hours
  Time from the end of material preparation to a successful catheterisation.
evaluate rescue technique | Up to 4 hours
  Rescue system chosen by the carer after an initial failure (call a colleague, continue with the conventional method, ultrasound-guided technique, infrared illumination technique or abandon peripheral venous insertion).
Evaluate Catheter size | Up to 4 hours
  Catheter sizes chosen by carers

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers Hospital, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol